CLINICAL TRIAL: NCT02775760
Title: The Entorhinal Cortex and Aerobic Exercise in Aging
Acronym: ECE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended due to Covid-19 policies, then terminated.
Sponsor: Boston University (Other)
Collaborators: Brigham and Women's Hospital (Other); Georgia Institute of Technology (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-34579; R21AG049968 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging
Keywords: brain; brain mapping; cognition; exercise; physical activity; hippocampus; entorhinal cortex; spatial navigation; learning; memory; magnetic resonance imaging; functional neuroimaging; physical endurance; physical fitness; resistance training; walking; muscle stretching exercises; exercise test; neuropsychological tests; executive function; attention; body composition
MeSH Terms: conditions — Motor Activity; Spatial Navigation | interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiovascular endurance (Experimental): Participants will undergo cardiovascular endurance training. The trainer-supervised endurance training will involve walking on a treadmill at moderate intensity
  Interventions: Behavioral: Cardiovascular endurance
- Strength, balance, and flexibility (Active Comparator): Participants will undergo Strength, balance, and flexibility training.
  Interventions: Behavioral: Strength, balance, and flexibility

INTERVENTIONS:
Behavioral: Cardiovascular endurance — Physical exercise at the Boston University Fitness and Recreation Center
  Arms: Cardiovascular endurance
Behavioral: Strength, balance, and flexibility — Physical exercise at the Boston University Fitness and Recreation Center
  Arms: Strength, balance, and flexibility

SUMMARY:
The overall goal of this study is to examine how regular exercise affects brain function, spatial memory, and virtual navigation. Participation in this research study will take approximately 4 months.

DETAILED DESCRIPTION:
The investigators are examining the effects of exercise and cardiovascular fitness on cognitive processes. Specifically, the investigators are examining if exercise improves brain function in a brain area known as the entorhinal cortex. Together with the hippocampus this brain area is important for memory formation and spatial navigation. Participation in this research study will take approximately 4 months. During this time, participants will make three initial study visits. The first visit is for informed consent and screening, the second visit is for baseline fitness testing, and the third visit is for cognitive testing and a functional MRI exam. Functional MRI is a brain imaging technique that uses a magnetic field to "take pictures" of the brain while a person performs a cognitive task. It will take up to approximately three weeks to complete these initial three study visits. Following the three initial study visits, the exercise-training program will begin. Participants will be randomized to one of two training programs: a cardiovascular endurance-training program (aerobic exercise) and a strength, balance, and flexibility training program (non-aerobic exercise). The exercise training program will last 12 weeks. There will be three one-hour exercise sessions per week. After completion of the exercise-training program, participants will attend two follow-up study visits. The first follow-up visit is for fitness testing. The second follow-up visit is for cognitive testing and an MRI exam.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-80 years
* Physical inactivity/sedentary status (The American College of Sports Medicine defines a sedentary lifestyle as a lifestyle in which a person is not participating in at least 30 minutes of moderate intensity physical activity on at least three days per week for at least three months.)
* Generally healthy
* Living in the greater Boston area
* Fluent in English (must have attended elementary school and higher in English)
* Non-smoking

Exclusion Criteria:

* Poor vision that cannot be corrected with glasses or contact lenses
* Presence of an acute infection
* Diagnosis of kidney failure
* Diagnosis of liver disease
* Diagnosis of thyrotoxicosis/hyperthyroidism
* Diagnosis of cancer
* Diagnosis of severe anemia
* Past or present conditions that affect cognitive functioning:

  * learning disability
  * neurological disorders or conditions (movement disorder, history of head trauma or stroke, epilepsy, etc.)
  * psychiatric disorders or conditions within last 5 years (depression, anxiety disorder, etc.)
  * Severe stress
* Evidence of cognitive impairment (e.g. dementia)
* Claustrophobia (fear of small, enclosed spaces)
* Obesity
* Past or present conditions that are counter indicators for participation in cardio-respiratory fitness assessment and physical exercise:

  * heart conditions (e.g. heart attack, arrhythmias, etc.)
  * circulatory conditions (e.g. uncontrolled hypertension, leg claudication, high cholesterol, etc.)
  * respiratory conditions (e.g., asthma or lung conditions, such as chronic obstructive pulmonary disease, acute bronchitis, acute common cold, lung cancer, pneumonia, etc.)
  * current musculoskeletal impairments (e.g. fractures, hemiplegia, chronic joint pain, arthritis, osteoporosis, not able to walk comfortably without assistance, etc.)
  * diagnosis of electrolyte disorder or abnormality
  * presence of diabetes mellitus
* Prescription medication or other drugs that treat heart, lung, or circulatory conditions (e.g. beta blockers, bronchodilators, etc.)
* Prescription medication or other drugs that affect chemicals in the brain (e.g. antidepressants, anxiolytics, etc.)
* Drug abuse or alcohol misuse
* Metal in or on the body that cannot be removed (e.g. pacemaker, defibrillator, metal implant that is ferrous)
* Some known abnormal MRI findings (case by case basis)
* Regularly exercising
* Unavailable for the approx. 4-month duration of the study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Schon, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kern KL, Storer TW, Schon K. Cardiorespiratory fitness, hippocampal subfield volumes, and mnemonic discrimination task performance in aging. Hum Brain Mapp. 2021 Mar;42(4):871-892. doi: 10.1002/hbm.25259. Epub 2020 Dec 16. PMID 33325614
- See also: Brain Plasticity and Neuroimaging Laboratory at Boston University — http://sites.bu.edu/brainplasticity/contact-us/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were first pre-screened over the telephone. At their initial visit, they gave written informed consent for all study procedures (screening, MRI, etc.). Thus, we consider every participant as enrolled who provided consent, and the number of participants started is not the same as the number of participants who were assigned to each Arm. 8 enrolled participants did not start the exercise intervention, 21 were not eligible after screening, leaving 29 who started the intervention.
Period: Overall Study
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Started | 17 | 12
Completed | 12 | 7
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 13 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.94 (5.40) | 68.75 (5.77) | 68.86 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Functional MRI - Right Subiculum
Description: The fMRI is measuring blood oxygenation levels and blood flow in different regions of the brain and using that to determine activity changes in the brain. This measurement was obtained while participants were performing a virtual navigation task in the MRI scanner.
  Data reported for fMRI is in beta-weight for navigation greater control contrast of BOLD images. The beta-weight is a standardized regression coefficient. Higher beta-weights mean greater activation and lower beta-weights mean less activation in specific brain regions being monitored. Negative beta-weights mean lower activation for the navigation condition than for the control condition, positive beta-weights mean greater activation for the navigation condition than for the control condition.
Time Frame: 0 months-baseline (pre-intervention)
Population: 3 participants were excluded due to excess head motion during functional MRI (2 RT, 1 ET), 1 participant was excluded because this participant did not complete the post-intervention MRI (1 ET) (ET = endurance training, RT = resistance training)
Measure: Mean (Standard Deviation); unit: BOLD Signal (beta weight)
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 10 | 5
BOLD Signal (beta weight) | -0.07876229 (0.233351521) | -0.14511014 (0.141012355)

2. Primary Outcome: Structural MRI - Right Dentate Gyrus Head
Description: Measurement of regional brain volumes in the medial temporal lobes to assess change in regional brain volumes. Reported outcome measure is volume of the right anterior (i.e., head) dentate gyrus, a hippocampal subfield known to show plasticity in response to exercise in animal models. The hippocampus is part of the medial temporal lobes.
Time Frame: 0 months-baseline (pre-intervention)
Population: 1 participant was excluded because this participant did not complete the post-intervention MRI (1 ET) (ET = endurance training)
Measure: Mean (Standard Deviation); unit: volume in cubic mm
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 11 | 7
volume in cubic mm | 142.7478413 (14.36877697) | 137.1801957 (19.71149913)

3. Primary Outcome: Cognitive Test Performance: Spatial Memory
Description: Participants will perform a spatial memory test during functional MRI. Measurements include baseline-to-follow-up change test performance.
Time Frame: 4 months
Population: Data not analyzed due to technical errors with the virtual reality (VR) navigation software platform.
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Cognitive Test Performance: Virtual Navigation
Description: Participants will perform a virtual navigation test during functional MRI. Measurements include baseline-to-follow-up change in test performance.
Time Frame: 4 months
Population: Data not analyzed due to technical errors with the virtual reality (VR) navigation software platform.
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Functional MRI - Post-intervention Right Subiculum
Description: as for outcome 1
Time Frame: 4 months
Population: 3 participants were excluded due to excess head motion during fMRI (2 RT, 1 ET), 1 participant was excluded because this participant did not complete the post-intervention MRI (1 ET) (ET = endurance training, RT = resistance training)
Measure: Mean (Standard Deviation); unit: BOLD Signal (beta weight)
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 10 | 5
BOLD Signal (beta weight) | 0.00078057 (0.242816203) | -0.17106976 (0.231649625)

6. Primary Outcome: Structural MRI - Post-intervention Right Dentate Gyrus Head
Description: as for outcome 2
Time Frame: 4 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: volume in cubic mm
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 11 | 7
volume in cubic mm | 143.0254936 (16.36761426) | 134.9353733 (23.23778171)

7. Secondary Outcome: Aerobic Capacity
Description: Participants will perform a treadmill test to estimate baseline-to-follow-up change in aerobic capacity. Aerobic capacity is the maximum amount of oxygen (O2;(expressed in volume: VO2) a person can utilize during strenuous exercise. This maximum volume of oxygen is known as VO2max or aerobic capacity. For this study, we measured heart rate during the treadmill test and estimated VO2max from heart rate, thus we estimated VO2max rather than measured oxygen and carbondioxyde in the breath while exercising. VO2max is expressed in milliliters per kilogram of body weight per minute (ml/kg/min). We calculated percentage change from baseline to post-intervention.
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Groups:
- Cardiovascular Endurance: Participants will undergo cardiovascular endurance training. The trainer-supervised endurance training will involve walking on a treadmill at moderate intensity Cardiovascular endurance: Physical exercise at theBoston University Fitness and Recreation Center
- Strength, Balance, and Flexibility: Participants will undergo Strength, balance, and flexibility training. Strength, balance, and flexibility: Physical exercise at the Boston University Fitness and Recreation Center
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 12 | 7
Percentage change from baseline | 18.32 [11.63 to 20.56] | 2.62 [1.22 to 16.12]

8. Secondary Outcome: Muscle Strength
Description: Participants will perform several muscle strength tests to estimate baseline-to-follow-up change in muscle strength. Percentage change in chess press weight lifted is reported in results.
Time Frame: 4 months
Population: All participants who completed the intervention were included in the analysis (12 cardiovascular endurance group, 7 strength, balance, and flexibility group).
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
Number analyzed (Participants) | 12 | 7
Percentage change from baseline | 0 [-8.75 to 13.92] | 17.24 [12.55 to 27.86]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Cardiovascular Endurance | Strength, Balance, and Flexibility
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/12
Other Adverse Events (participants affected / at risk) | 3/17 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cardiovascular Endurance (N=17) | Strength, Balance, and Flexibility (N=12)
Fainting (Gastrointestinal disorders) | 0 | 1 — 1 participant reported being admitted to an emergency department due to fainting spells
Sciatica pain (Nervous system disorders) | 1 | 0
Sudden tachycardia (Cardiac disorders) | 1 | 0 — Participant was subsequently diagnosed with atrial fibrillation (no hospitalization needed), and participation was terminated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cardiovascular Endurance (N=17) | Strength, Balance, and Flexibility (N=12)
hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Concussion (Nervous system disorders) | 0 | 1 — Unrelated to research study (due to accident that happened at participant's home)
Back soreness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 — right foot
Headache (Nervous system disorders) | 0 | 1
tachycardia and chest tightness (Cardiac disorders) | 1 | 0 — EMT suspected heart rate monitor dysfunction and a subsequent panic attack

LIMITATIONS AND CAVEATS:
Note the small number of participants with complete pre- and post-intervention datasets (N=19). This number was even lower for functional MRI data analyses due to excessive head motion. This limits the interpretation of the results. In addition, the trial was also suspended and then terminated due to the SARS-CoV-2 (COVID-19) pandemic, which also contributed to data loss.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT02775760/Prot_SAP_000.pdf